CLINICAL TRIAL: NCT04195009
Title: Observational Study Evaluating the Impact of Surgical Stress Suppression During Opioid Free Anesthesia on Postoperative Inflammation During Major Surgery.
Brief Title: Impact of Suppressing Surgical Stress Reaction on Postoperative Inflammation.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Principal investigator, AZ Sint-Jan AV
Other Study IDs: OS impact SSR on SIRS d OFA
Record Dates: First submitted 2019-12-02; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Inflammation; Postoperative Pain
MeSH Terms: conditions — Inflammation; Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: major surgery under opioid free anesthesia without regional anesthesia — measuring nociception in every patient but blinded for attending anesthesiologist

SUMMARY:
Patients undergoing surgery under opioid free general anesthesia (OFA) are monitored with antinociceptive devices like NOL or ANI that measures sympathetic activity but are invisible for the attending anesthesiologist . Observational study comparing patients with sufficient suppression of sympathetic reactions with patients having insufficient suppression on hemodynamic stability, post operative sedation, pain and inflammatory markers.

DETAILED DESCRIPTION:
all patients get an opioid free anesthesia using dexmedetomidine, lidocaine, ketamine and magnesium. dosing is according to the attending anesthesiologist.

total dose of each drug and duration of anesthesia are recorded. Antinociceptive devices measures how long the patient is during anesthesia having a nociceptive level nociception level index (NOL) or Analgesia Nociception Index (ANI) above normal without showing the data to the attending anesthesiologist.

Relationship is calculated between on one side the hemodynamic stability, postoperative sedation, pain, postoperative CRP and on the other side the time NOL is above 20 or ANI is below 50.

ELIGIBILITY:
Inclusion Criteria:

* major surgical procedures without need for regional anesthesia

Exclusion Criteria:

* allergy to one of the anesthetics used
* major liver, renal cardiac or pulmonary disease reducing normal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major surgical procedures without need for regional anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
CRP 24 hours postoperative | 24 hours postoperative
  measure chronic reactive protein (CRP) biomarker of surgical inflammation

SECONDARY OUTCOMES:
hemodynamic stability | intraoperative
  dosis of vasoactive drugs needed to support blood pressure before blood pressure rise as requested by surgeons.
postoperative pain using VAS score | up to 4 hours postoperative during post anesthetic care unit (PACU) stay
  postoperative pain measured by visual analog scale (VAS) score: max pain =10 and worst, no pain = 0
postoperative sedation using Ramsay score | first 4 hours postoperative during PACU stay
  deepest postoperative sedation level measured by the Ramsay score at the PACU full awake or no sedation = 1 deep sleep or anesthesia = 5 and worst
postoperative opioids used | first 24 hours postoperative
  total amount of opioids needed postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, MD PhD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No